CLINICAL TRIAL: NCT02010853
Title: Transient Global Amnesia (TGA) Exploratory Study of the Default Mode Network in Resting State Functional MRI (fMRI) During the Acute Phase
Brief Title: Transient Global Amnesia (TGA). Exploratory Study of the Default Mode Network During the Acute Phase
Acronym: ICTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13 201 02; 2013-A01271-44 (Other: ANSM -IDRCB)
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Amnesia
Keywords: Transient Global amnesia; fMRI; resting state
MeSH Terms: conditions — Amnesia; Amnesia, Transient Global

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient (Experimental): each patient TGA will receive an evaluation in resting state IRMf during three successive visits:
  * During the acute phase within 24 hours
  * In 72 hours
  * In 3 months
  Interventions: Other: IRMf
- control (Other): each control will receive an evaluation in resting state IRMf during three successive visits:
  * During the acute phase within 24 hours
  * In 72 hours
  * In 3 months
  Interventions: Other: IRMf

INTERVENTIONS:
Other: IRMf — evaluation in resting state fMRI during three successive visits:
  * During the acute phase within 24 hours
  * In 72 hours
  * In 3 months

SUMMARY:
The transient global amnesia, in which the memory disorder is massive, transient and pure, offers a unique model for exploring episodic memory. Topographic MRI can reveal a focal and selective lesion located on the CA1 region of the hippocampus better visible between 48h and 72h after onset of the episode.

There is therefore a real dissociation between structural lesions witch are minimal or non-existent and the massive memory disorder. This suggests that functional impairment goes far beyond the structural damage in this condition. To our knowledge, no study has been performed to identify this functional impairment using resting state fMRI.

Thus, investigators wish to study the neural networks involved in memory impairment during the acute phase of transient global amnesia using resting state imaging. This technique appears to be modern and adapted to these patients population. Investigators hypothesize that despite limited structural lesions, a large functional network is impaired compared to that observed in a group of healthy subjects. investigators believe that the alteration of the functional network will explain the depth of memory impairment observed.

The main aim of this study will be to identify functional impairment in the patient group vs. control group during the acute phase of transient global amnesia (TGA) using resting state imaging.

Patients potentially eligible will be informed during their arrival to the emergency unit. If the patient is eligible and would like to participate, information will be given. For the patients willing to participate, inclusion and exclusion criteria will be verified. Two imaging exams (topographic MRI and resting state fMRI) and neuropsychological assessment will be performed during three visits.

DETAILED DESCRIPTION:
Background:

The transient global amnesia is a transient, massive and pure memory disorder. Its pathophysiology is poorly known, but the disease process involves the Papez circuitry, and more specifically the medial part of the temporal lobes (hippocampi). It involves 3-8 per 100,000 people per year. The age of patients affected is between 50 and 70 years. Structural MRI can confirm the diagnosis by revealing a focal and selective lesion located on the CA1 region of the hippocampus better observed between 48h and 72h after onset of the episode.

Main purpose:

The main aim of this study is to identify neuronal functional impairment in a group of patients vs. a group of healthy subjects during the acute phase of transient global amnesia (TGA) using resting state fMRI imaging.

Secondary purpose:

* Show correlations between functional activity observed in resting state fMRI at the acute phase and cognitive performance in the patient group.
* Describe the evolution of functional impairment in resting state fMRI between the acute phase (visit 1) and post-acute phases (visit 2 and 3) in the patient group compared to the control group subjects.

Study design:

Monocentric, pilot, prospective, controlled study including consecutive patients admitted to the emergency department of the CHU of Toulouse for transient global amnesia. investigators will compare two independent groups: patients and controls We expect three months between the signing of consent and the end of the study. The total duration of the study will not exceed 27 months.

Arm number or label and arm type: This study is exploratory. investigators will compare two independent groups: patients and controls

Interventions:

After signing the informed consent each patient TGA will receive a neuropsychological assessment, a topographic MRI and an evaluation in resting state fMRI during three successive visits:

* During the acute phase within 24 hours
* In 72 hours
* In 3 months

Number of subjects:

It's difficult to estimate the number of subjects required to show a difference in resting state between the two groups during the acute phase of TGA. No study of that type in the literature is available to estimate the sample size to be recruited. In this pilot study we will recruit 22 subjects in each group.

Expected benefits:

The transient global amnesia is a model for exploring memory because this disorder is massive, pure and temporary. Better understand the Neural Network substrates underlying this alteration could help to better understand memory disorders in other diseases (Korsakoff syndrome, thalamic stroke, dissociative amnesia, Alzheimer's disease). Such discovery could lead to clinical trials of functional brain stimulation as recently developed in other neurological disorders in which functional impairment has been shown. (TMS, TDCS)

Statistical analysis:

The SPM8 software will be used to generate activation map using fMRI images. The obtained maps will be compared between groups using t test imbedded in the same software. Correlation maps between cognitive performance and activation will be also calculated. Intra group comparison across time will then be assessed.

ELIGIBILITY:
Inclusion Criteria:

Patient group

Clinical criteria of definition of transient global amnesia:

Acute disorder of anterograde memory observed by a witness. Respect of the other cognitive functions. No exclusion criteria for this diagnosis (see exclusion criteria section).

Hippocampal lesion in DWI MRI performed at 72h Clinical resolution of memory disorder within 24 hours

Control group No cognitive complaint No history of transient amnesia

Both groups Age between 40 and 80 years old

Exclusion Criteria:

Patient group Disturbance of consciousness or loss of identity Argument in favor of seizure disorders Presence of a neurological deficit focused

Both groups Recent head trauma Acute intoxication ethyl Taking drugs influencing memory processing Severe hypoglycemia Psychiatric disorder altering capacity for judgment Progressive neurological disorder with cognitive alteration Indication against MRI French language level insufficient to be appropriately involved in neuropsychological assessment, Administrative issues: unable to give informed about information, not covered by a social security system, refusal to sign the consent, patient under curators.

Pregnant Woman

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The primary judgment criteria will be the difference in activation probabilistic resting state maps between patient and control groups during the acute phase. | 3 months

SECONDARY OUTCOMES:
memory performance tests and functional activity | 3 months
  The correlation coefficient between memory performance tests and functional activity observed in resting state fMRI in the group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: PrJérémie Pariente, PHD, Principal Investigator — Department of Neurology, Purpan Hospital, Toulouse
Locations (1):
- Chu Purpan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No